CLINICAL TRIAL: NCT00771810
Title: Ph IIb Study Evaluating the Safety & Efficacy of TXA127 in the Reduction of Incidence and Severity of Thrombocytopenia in Patients Receiving Combination Gemcitabine and Platinum Therapy for Ovarian, Fallopian Tube, or Peritoneal Carcinoma
Brief Title: Study of Drug to Reduce Thrombocytopenia in Patients Receiving Chemo for Ovarian, Fallopian Tube or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tarix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TXA127-2007-002
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Results first posted 2013-06-07 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Thrombocytopenia; Neutropenia; Lymphopenia; Anemia
Keywords: Ovarian Cancer; Thrombocytopenia; Cytopenia; Chemotherapy
MeSH Terms: conditions — Thrombocytopenia; Neutropenia; Lymphopenia; Anemia; Ovarian Neoplasms; Cytopenia | interventions — angiotensin I (1-7)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Combination gemcitabine and platinum-based chemotherapy with concurrent placebo
  Interventions: Drug: Placebo
- TXA127 100 ug/kg (Experimental): Combination gemcitabine and platinum-based chemotherapy with concurrent 100 ug/kg/day TXA127
  Interventions: Drug: TXA127
- TXA127 300 ug/kg (Experimental): Combination gemcitabine and platinum-based chemotherapy with concurrent 300 ug/kg/day TXA127
  Interventions: Drug: TXA127

INTERVENTIONS:
Drug: TXA127 — Once daily subcutaneous injection of 100 ug/kg
  Other Names: Angiotensin 1-7
  Arms: TXA127 100 ug/kg
Drug: TXA127 — Once daily subcutaneous injection of 300 ug/kg
  Other Names: Angiotensin 1-7
  Arms: TXA127 300 ug/kg
Drug: Placebo — Once daily subcutaneous injection of placebo
  Arms: Placebo

SUMMARY:
This research study will investigate the safety and effectiveness of two different dose levels of a new, unapproved drug to be given along with the chemotherapy regimens gemcitabine and carboplatin or gemcitabine and cisplatin prescribed to women for the treatment of ovarian cancer. This experimental drug is called TXA127 and is being tested for effectiveness to see if it will help reduce some of the side effects of the chemotherapy, primarily low blood platelet levels that lead to excess bleeding. This study also intends to test the safety of TXA127 when given as an injection under the skin on a daily basis concurrently with up to 6 cycles of the prescribed chemotherapy.

DETAILED DESCRIPTION:
This is a Phase IIb, multicenter, randomized, double-blind, placebo-controlled study comparing safety and efficacy of two dose levels of TXA127 when administered during 6 cycles of combination gemcitabine and platinum-based chemotherapy. This study intends to investigate the effectiveness of TXA127 for the mitigation of severity and/or incidence of thrombocytopenia, as well as safety when administered as a self-injected, subcutaneous solution.

Females 18 years of age or older with a confirmed diagnosis of ovarian carcinoma who are scheduled to undergo combination chemotherapy with gemcitabine and carboplatin or gemcitabine and cisplatin will be considered for this study. Subjects may be chemotherapy naïve, newly diagnosed, or post a single course of chemotherapy followed by a progression- and treatment-free interval of at least 3 months, or post 2 or more previous courses of chemotherapy after a progression- and treatment-free interval of at least 6 months.

Subjects will be randomized in a 1:1:1 ratio to one of the following three blinded treatment groups: placebo, 100 ug/kg/day TXA127 and 300 ug/kg/day TXA127.

Treatment will be concurrent with up to six consecutive 21-day cycles of one of the following gemcitabine and platin regimens:

Regimen A

* Intravenous cisplatin therapy at a dose of 30-50 mg/m2 given on Day 1 of the cycle
* Intravenous gemcitabine at a dose of 800 mg/m2 given on Day 1 after cisplatin and on Day 8 of the cycle.

Regimen B

* Intravenous gemcitabine at a dose of 1000 mg/m2 given on Days 1 and 8 of the cycle
* Intravenous carboplatin AUC 4 given after gemcitabine on Day 1 of the cycle

TXA127 will be self-administered as a subcutaneous injection by the subject once daily on Days 2-6 and 9-15 during each cycle of chemotherapy. Blood specimens will be drawn for hematologic analysis on Days 1, 8 and 15 of each treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Females at least 18 years of age with ovarian carcinoma who are one of the following:

  * Newly diagnosed with ovarian cancer and chemotherapy naïve, or
  * Post a single previous course of chemotherapy, with a 3-month disease-progression and treatment-free interval, with the exception of antibody therapy, prior to the study screening visit, or
  * Post two or more previous courses of chemotherapy with a 6-month disease-progression and treatment-free interval, with the exception of antibody therapy, prior to the study screening visit.
* Must be scheduled for a course of combination chemotherapy consisting of gemcitabine and cisplatin or gemcitabine and carboplatin to be administered in 21-day cycles
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Adequate bone marrow, renal, and hepatic functions as measured by standard chemistry and hematology blood tests
* Adequate blood coagulation parameters as measured by standard blood tests for coagulation

Exclusion Criteria:

* Any clinical or laboratory abnormality greater than Grade 2 toxicity (NCI criteria), with the exception of laboratory parameters specified in the inclusion criteria
* Significant unstable cardiovascular disease
* Uncontrolled high blood pressure
* Current use of an angiotensin converting enzyme (ACE) inhibitor or angiotensin II antagonists
* Evidence of metastatic disease to the bone
* Metastatic disease to the CNS requiring treatment or radiation therapy
* Uncontrolled infection(s)
* Radiation therapy or chemotherapy (except as specified in the inclusion criteria) within the previous 5 years
* Concurrent use of hematopoietic or erythropoietic agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gere S diZerega, MD, Study Director — US Biotest, Inc.
Locations (6):
- United States (6):
  - University of Southern Alabama Mitchell Cancer Institute, Mobile, Alabama
  - USC - LAC Medical Center, Los Angeles, California
  - University of California - Irvine, Chao Family Comprehensive Cancer Center, Orange, California
  - Rush University Medical Center, Chicago, Illinois
  - Associates in Women's Health, Wichita, Kansas
  - Schwartz Gynecologic Oncology, PLLC, Brightwaters, New York

REFERENCES:
- [Background] Rodgers KE, Oliver J, diZerega GS. Phase I/II dose escalation study of angiotensin 1-7 [A(1-7)] administered before and after chemotherapy in patients with newly diagnosed breast cancer. Cancer Chemother Pharmacol. 2006 May;57(5):559-68. doi: 10.1007/s00280-005-0078-4. Epub 2005 Aug 12. PMID 16096787
- [Background] Ellefson DD, diZerega GS, Espinoza T, Roda N, Maldonado S, Rodgers KE. Synergistic effects of co-administration of angiotensin 1-7 and Neupogen on hematopoietic recovery in mice. Cancer Chemother Pharmacol. 2004 Jan;53(1):15-24. doi: 10.1007/s00280-003-0710-0. Epub 2003 Oct 16. PMID 14569417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Feb2009 to Feb2012 across 10 oncology sites.
Groups:
- Placebo: Group 1: combination gemcitabine and platinum-based chemotherapy with concurrent placebo
- TXA127 100 ug/kg: Group 2: combination gemcitabine and platinum-based chemotherapy with concurrent 100 ug/kg/day TXA127
- TXA127 300 ug/kg: Group 3: combination gemcitabine and platinum-based chemotherapy with concurrent 300 ug/kg/day TXA127
Period: Overall Study
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300 ug/kg
Started | 10 | 11 | 13
Completed | 5 | 6 | 6
Not Completed | 5 | 5 | 7
Not completed — Adverse Event | 3 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 1 | 2 | 2
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TXA127 300ug/kg: Group 3: combination gemcitabine and platinum-based chemotherapy with concurrent 300 ug/kg/day TXA127
- Total: Total of all reporting groups
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300ug/kg | Total
Number analyzed (Participants) | 10 | 11 | 13 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 10 | 27
  >=65 years | 2 | 2 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 13 | 34
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 11 | 13 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 8 | 9 | 11 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 13 | 34

OUTCOME MEASURES:

1. Primary Outcome: Chemotherapy Cycles During Which the Platelet Count Measures Below 50,000/mm3
Description: Mean percentage of cycles with platelet counts below 50,000/mm3
Time Frame: During a maximum of six 3-week chemotherapy cycles
Population: The number of participants for analysis was the intention to treat population.
Measure: Mean (Full Range); unit: Percentage of cycles
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300ug/kg
Number analyzed (Participants) | 10 | 10 | 12
Percentage of cycles | 20.0 [0 to 67] | 11.7 [0 to 50] | 21.5 [0 to 100]

2. Secondary Outcome: Subjects With Platelet Counts Below 50,000/mm3
Description: Number of subjects who experienced a platelet count below 50,000/mm3
Time Frame: During a maximum of six 3-week chemotherapy cycles
Population: The number of participants for analysis was the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300ug/kg
Number analyzed (Participants) | 10 | 11 | 13
Participants | 5 | 4 | 6

3. Secondary Outcome: Treatment Cycles With Platelets Counts Below 25,000/mm3
Description: Mean percentage of treatment cycles where platelets counts were below 25,000/mm3
Time Frame: During a maximum of six 3-week chemotherapy cycles
Population: The number of participants for analysis was the intention to treat population.
Measure: Mean (Full Range); unit: Percentage of cycles
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300ug/kg
Number analyzed (Participants) | 10 | 10 | 12
Percentage of cycles | 5.8 [0 to 33.3] | 0 [0 to 0] | 10.4 [0 to 83.3]

4. Secondary Outcome: Chemotherapy Dose Intensity and Dose Density
Description: Mean percentage of cycles where projected (target) chemotherapy dose was maintained
Time Frame: During a maximum of six 3-week chemotherapy cycles
Population: The number of participants for analysis was the intention to treat population.
Measure: Mean (Full Range); unit: Percentage of cycles
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300ug/kg
Number analyzed (Participants) | 10 | 10 | 12
Percentage of cycles
  Gemcitabine | 67.6 [46.3 to 100.0] | 86.5 [61.4 to 102.3] | 71.7 [45.0 to 95.5]
  Gemcitabine with Carboplatin or Cisplatin | 76.7 [59.8 to 100.0] | 88.7 [68.0 to 99.1] | 79.5 [51.4 to 96.3]

5. Secondary Outcome: Lymphopenia as Determined by Lymphocyte Count
Description: Number of subjects with a treatment emergent adverse event of lymphopenia
Time Frame: During a maximum of six 3-week chemotherapy cycles
Population: The number of participants for analysis was the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300 ug/kg
Number analyzed (Participants) | 10 | 11 | 13
Participants | 1 | 0 | 0

6. Secondary Outcome: Neutropenia
Description: Number of subjects with a treatment emergent adverse event of neutropenia
Time Frame: During a maximum of six 3-week chemotherapy cycles
Population: The number of participants for analysis was the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300 ug/kg
Number analyzed (Participants) | 10 | 11 | 13
Participants | 7 | 5 | 8

7. Secondary Outcome: Anemia
Description: Number of subjects with a treatment emergent adverse event of anemia
Time Frame: During a maximum of six 3-week chemotherapy cycles
Population: The number of participants for analysis was the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300 ug/kg
Number analyzed (Participants) | 10 | 11 | 13
Participants | 2 | 4 | 5

8. Secondary Outcome: Mucositis
Description: Number of subjects with a treatment emergent adverse event of mucositis
Time Frame: During a maximum of six 3-week chemotherapy cycles
Population: The number of participants for analysis was the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300 ug/kg
Number analyzed (Participants) | 10 | 11 | 13
Participants | 2 | 0 | 1

9. Secondary Outcome: Alopecia
Description: Number of subjects with a treatment emergent adverse event of alopecia
Time Frame: During a maximum of six 3-week chemotherapy cycles
Population: The number of participants for analysis was the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300 ug/kg
Number analyzed (Participants) | 10 | 11 | 13
Participants | 1 | 2 | 3

10. Secondary Outcome: Rescue Treatment for Hematopoiesis and Mucositis
Description: Number of subjects with a treatment emergent adverse event of hematopoiesis and mucositis who received rescue treatment as determined by the administration of:
  1. Transfusions
  2. Filgrastim or Pegfilgrastim
  3. Erythropoietin
  4. Palifermin
Time Frame: During a maximum of six 3-week chemotherapy cycles
Population: The number of participants for analysis was the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300 ug/kg
Number analyzed (Participants) | 10 | 11 | 13
Participants
  Hematopoiesis - Transfusions | 2 | 4 | 2
  Hematopoiesis - Filgrastim or Pegfilgrastim | 4 | 2 | 5
  Hematopoiesis - Erythropoietin | 0 | 0 | 0
  Mucositis - Palifermin | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: February 2009 to May 2011
Description: The assessment types were coded using MedDRA.
Arm/Group | Placebo | TXA127 100 ug/kg | TXA127 300 ug/kg
Serious Adverse Events (participants affected / at risk) | 3/10 | 1/11 | 3/13
Other Adverse Events (participants affected / at risk) | 10/10 | 11/11 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | TXA127 100 ug/kg (N=11) | TXA127 300 ug/kg (N=13)
Abdonminal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Female genital tract fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion with dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | TXA127 100 ug/kg (N=11) | TXA127 300 ug/kg (N=13)
Anaemia (Blood and lymphatic system disorders) | 2 (8) | 4 (16) | 5 (10)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (13) | 3 (3) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (21) | 5 (13) | 8 (18)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (10) | 5 (15) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Ascites (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Cardiac disorders) | 3 (5) | 3 (10) | 3 (11)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (7)
Abdominal pain (Gastrointestinal disorders) | 5 (9) | 4 (4) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ageusia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (10) | 7 (12) | 5 (9)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 1 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Female genital tract fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (18) | 7 (17) | 9 (16)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Pharyngitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1)
Tooth abscess (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (7) | 4 (9) | 5 (6)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 2 (5)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (2) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (2) | 1 (2) | 1 (1)
Device leakage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device related infection (General disorders) | 0 (0) | 0 (0) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 8 (12) | 6 (17) | 7 (23)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 3 (3)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hot flush (General disorders) | 2 (2) | 0 (0) | 0 (0)
Incision site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Induration (General disorders) | 1 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (6) | 2 (2) | 2 (2)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (General disorders) | 2 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 2 (2) | 2 (8)
Pain (General disorders) | 1 (1) | 2 (2) | 3 (14)
Postoperative fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 3 (8) | 2 (2)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 5 (6) | 1 (1) | 2 (4)
Infusion related reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (4)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (16)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Transaminases abnormal (Investigations) | 0 (0) | 0 (0) | 1 (3)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Thirst (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (7) | 5 (8)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Chills (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 1 (1)
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (12) | 5 (8) | 5 (16)
Hypoaesthesia (Nervous system disorders) | 2 (3) | 0 (0) | 3 (5)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Tremors (Nervous system disorders) | 0 (0) | 0 (0) | 1 (4)
Urinary incontinence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0)
Crying (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 2 (3) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 2 (3) | 1 (2)
Enterovesical fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (3) | 1 (3) | 1 (1)
Urogenital fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Vaginal disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal lesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 5 (16)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Hair disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 5 (12)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin sensitisation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin warm (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Vascular disorders) | 3 (4) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (3) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Feasibility considerations (e.g., slow patient enrollment and lower incidence of Grade 3-4 thrombocytopenia than planned) necessitated early termination of the study after 34 patients had been enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days